CLINICAL TRIAL: NCT02838303
Title: The Use of Self-reported Symptoms as a Proxy for Acute Organophosphate Poisoning Among Nepali Farmers: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study
Brief Title: The Use of Self-reported Symptoms as a Proxy for Acute Organophosphate Poisoning Among Nepali Farmers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Augustinus Fonden (Other)
Responsible Party: Principal Investigator, Dea Haagensen Kofod, MB, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 12205-01-57-02
Record Dates: First submitted 2016-07-14; First posted 2016-07-20 (Estimated); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Organophosphate Poisoning
MeSH Terms: conditions — Organophosphate Poisoning | interventions — Organophosphates; Biological Control Agents

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Other): Initial spray session: organophosphate. Crossover spray session: placebo
  Interventions: Other: Organophosphate; Other: Placebo
- Group B (Other): Initial spray session: placebo. Crossover spray session: organophosphate
  Interventions: Other: Organophosphate; Other: Placebo

INTERVENTIONS:
Other: Organophosphate — Chlorpyrifos 50% plus cypermethrin 5%, WHO Class II: Moderately hazardous
Other: Placebo — Multineem, WHO Class U: Unlikely to present acute hazard in normal use
  Other Names: Biopesticide

SUMMARY:
The purpose of this study is to evaluate self-reported symptoms as a proxy for acute organophosphate poisoning by examining self-reported acute organophosphate poisoning symptoms and PchE activity in response to occupational acute organophosphate exposure among farmers in Nepal.

ELIGIBILITY:
Inclusion Criteria:

* male
* minimum age 18 years
* hand pressured backpack sprayer usage
* used to spray with moderately to extremely hazardous pesticides according to the World Health Organization's (WHO) Pesticide Hazard Classification

Exclusion Criteria:

* usual personal protective equipment use (respirator/mask with particulate filter, face shield, googles, gloves, boots, plastic poncho)
* unwilling to stay pesticide-free seven days prior to each of the two spray sessions
* medical conditions interfering with PchE activity (liver disease, acute infection, chronic malnutrition, heart attack, cancer, obstructive jaundice, inflammation caused by various diseases, or use of pyridostigmine drugs)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-09; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change in self-reported acute organophosphate poisoning symptoms from baseline to follow up | Obtained just before (baseline) and 30 minutes after (baseline) each spray session
  Obtained using a structured questionnaire interview. The definition of symptoms was based on WHO's standardized list of clinical presentations of acute organophosphate poisoning.
Change in Plasma Cholinesterase (PchE) activity from baseline to follow up | Obtained just before (baseline) and 30 minutes after (baseline) each spray session
  PchE activity was measured with a blood test using a Test-mate Che Cholinesterase System (Model 400) with a PchE Plasma Cholinesterase Assay Kit (Model 470).

CONTACTS AND LOCATIONS:
Overall Officials: Dea H. Kofod, MB, Principal Investigator — Department of Occupational and Environmental Medicine, Bispebjerg Frederiksberg Hospital, University of Copenhagen

REFERENCES:
- [Derived] Kofod DH, Jors E, Varma A, Bhatta S, Thomsen JF. The use of self-reported symptoms as a proxy for acute organophosphate poisoning after exposure to chlorpyrifos 50% plus cypermethrin 5% among Nepali farmers: a randomized, double-blind, placebo-controlled, crossover study. Environ Health. 2016 Dec 13;15(1):122. doi: 10.1186/s12940-016-0205-1. PMID 27964728